CLINICAL TRIAL: NCT02699476
Title: Enhancing Cognitive and Neurobehavioral Functions After Repetitive Traumatic Brain Injuries (rTBI) in Retired NFL Players and Military Veterans.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brain & Body Health Foundation (Other)
Responsible Party: Principal Investigator, Robert W. Van Boven, M.D., D.D.S., Director, Brain & Body Health Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BBHF-001
Record Dates: First submitted 2016-02-26; First posted 2016-03-04 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Traumatic Brain Injury; Concussion; Mild Cognitive Disorder
Keywords: NFL; veterans; cognitive training; TBI; concussion
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion; Neurocognitive Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Individual + Computer A (Active Comparator): Daily activities involve playing one hour of computer games (e.g., hangman, boggle, word scramble, chess; computer cognitive training A (CCA)), and two (2) 90 minute individual training sessions interacting one-on-one with a trainer in a variety of cognitive tasks including attention, memory, and comprehension of information.
  Interventions: Behavioral: Interactive Trainer-Subject Sessions; Device: Active Control Games
- Individual + Computer B (Experimental): Daily activities involve playing an alternative set of computer games (computer cognitive training B (CCB)), and two (2) 90 minute individual training sessions interacting one-on-one with a trainer in a variety of cognitive tasks including attention, memory, and comprehension of information.
  Interventions: Device: Cognitive Behavioral Computer Training; Behavioral: Interactive Trainer-Subject Sessions
- Group + Computer B (Active Comparator): Daily activities involve group and individual cognitive therapy discussions on health, nutrition, and other topics and computer cognitive training B (CCB).
  Interventions: Behavioral: Psycho-Social Therapy; Device: Cognitive Behavioral Computer Training

INTERVENTIONS:
Behavioral: Psycho-Social Therapy
  Arms: Group + Computer B
Device: Cognitive Behavioral Computer Training
  Other Names: BrainHQ
  Arms: Group + Computer B; Individual + Computer B
Behavioral: Interactive Trainer-Subject Sessions
  Other Names: LearningRx
  Arms: Individual + Computer A; Individual + Computer B
Device: Active Control Games
  Arms: Individual + Computer A

SUMMARY:
The purpose of this study is to compare different combinations of cognitive training in retired professional football players and military veterans with a history of repeated concussions and persistent symptoms of impaired memory, concentration, attention, focus, or thinking.

ELIGIBILITY:
Inclusion Criteria:

* History of >1 Mild TBI: post traumatic amnesia/confusion ≤ 24 hour immediately after injury; or loss of consciousness <30 min confirmed by the Ohio State University TBI Identification Method-Short Form (OSU TBI-ID-SF).
* Age 25-55 years
* Minimum of 4 months post-injury
* Adequate visual, auditory, sensory-motor function for training program.
* Fluent in English
* Persistent cognitive dysfunction confirmed by Ruff Neurobehavioral Inventory score of greater than 70 on any of the four cognitive scales (Attention, Memory, Language, Executive).

Exclusion Criteria:

* History of hypoxic event
* Pre-existing significant neurological (e.g. MS) or psychiatric (e.g. schizophrenia, bi-polar) disorders.
* Current illicit drug use or alcohol abuse
* Unwilling or unable (e.g. language barrier) to participate
* Hospitalization during study
* Current Litigation
* Positive on malingering test
* Use of medications to enhance cognitive function (e.g. Ritalin)
* Initial Glasgow Coma Score < 13 or penetrating head injury
* Subjects must not show suicidal ideation as measured by the Columbia-Suicide Severity Rating Scale. Subjects with a score of 4 or 5 (as recommended by the FDA for treatment trials) will be excluded and referred for appropriate treatment.
* Subjects should not be enrolled in a concurrent TBI clinical trial.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Composite performance score based on battery of neuropsychological tests of working memory, learning, memory, and executive function. | within one week following treatment completion
  Composite performance score on neuropsychological battery based on four primary domains : learning, memory, working memory, and executive function.
Participant reported outcomes | within one week following treatment completion.
  Measure of impact of program use on the patient's own view of their impairment and function.
Working/school status | within one week following treatment completion.
  Measure of participants' employment status, and the number of hours worked/volunteered/in-school per week.
Exercise-base assessments | within one week following treatment completion.
  Four sets of assessments that are closely modeled on study-related exercises in the auditory, visual, cognitive, and social-cognitive modules. These include auditory speed of processing, visual speed of processing, cognitive control speed of processing and face recognition, recall of unique faces, and emotional cue recognition.
Functional assessments | within one week following treatment completion.
  Timed instrumental activities of daily living (TIADL) and the Mayo-Portland Adaptability Inventory (MPAI-4) for sensitive directly observed performance and well-accepted clinical impression measures.

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Van Boven, M.D., D.D.S., Principal Investigator — Brain & Body Health Foundation
Locations (1):
- Brain & Body Health Institute, P.A., Lakeway, Texas, United States

IPD SHARING:
Plan to Share IPD: No